CLINICAL TRIAL: NCT01244763
Title: A Phase 2, Randomized, Open-Label, Dose Titration, Efficacy and Safety Study of FG-4592 (Roxadustat) in Non-Dialysis Chronic Kidney Disease Patients With Anemia
Brief Title: Study of Roxadustat in Non-Dialysis Chronic Kidney Disease Participants With Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyntra Bio (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FGCL-4592-041
Record Dates: First submitted 2010-11-16; First posted 2010-11-19 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Chronic Kidney Disease; Anemia
Keywords: Kidney; Chronic Kidney Disease; CKD; Renal; Anemia; Oral anemia treatment; Hemoglobin levels; Erythropoietin; Blood count; Predialysis; Pre-dialysis; Hb; Non-dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort A: Roxadustat Tiered, Weight Based Dosing TIW (Experimental): Participants will receive roxadustat capsules, administered orally 3 times weekly (TIW) for 16 weeks. Initial roxadustat dose will be based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kilograms (kg)], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants will receive 60, 100, and 140 milligrams [mg] roxadustat, respectively). Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL.
  Interventions: Drug: Roxadustat
- Cohort B: Roxadustat Tiered, Weight Based Dosing TIW then BIW (Experimental): Participants will receive roxadustat capsules orally for 16 weeks. Initial roxadustat dose will be based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants will receive 60, 100, and 140 mg roxadustat, respectively). Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants will have a dose frequency reduction from TIW to 2 times a week (BIW) at the time of the initial Hb response.
  Interventions: Drug: Roxadustat
- Cohort C: Roxadustat at 50 mg TIW (Experimental): Participants will receive roxadustat capsules at 50 mg, administered orally TIW for 24 weeks. Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 10.5-12 g/dL.
  Interventions: Drug: Roxadustat
- Cohort D: Roxadustat at 100 mg TIW (Experimental): Participants will receive roxadustat capsules at 100 mg, administered orally TIW for 24 weeks. Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 10.5-12 g/dL.
  Interventions: Drug: Roxadustat
- Cohort E: Roxadustat Tiered, Weight Based Dosing BIW then QW (Experimental): Participants will receive roxadustat capsules for 24 weeks. Initial roxadustat dose will be based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants will receive 70, 100, and 150 mg roxadustat, respectively). Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.5 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants will have a dose frequency reduction from BIW to 1 time a week (QW) at the time of the initial Hb response.
  Interventions: Drug: Roxadustat
- Cohort F: Roxadustat at 70 mg BIW then QW (Experimental): Participants will receive roxadustat capsules at 70 mg for 24 weeks. Dose adjustments will be implemented (up to a maximum roxadustat dose of 2.5 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants will have a dose frequency reduction from TIW to BIW at the time of the initial Hb response. Then after >8 weeks of stable Hb, dose frequency will be reduced from BIW to QW.
  Interventions: Drug: Roxadustat

INTERVENTIONS:
Drug: Roxadustat — Oral capsule
  Other Names: FG-4592

SUMMARY:
The primary purpose of this study is to evaluate efficacy and safety of roxadustat in the correction of anemia in participants with non-dialysis chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Chronic kidney disease, not receiving dialysis
3. Body weight 45 to 140 kg

Exclusion Criteria:

1. Any clinically significant infection or evidence of an underlying infection
2. Positive for any of the following: human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibody (anti-HCV Ab)
3. History of chronic liver disease
4. New York Heart Association Class III or IV congestive heart failure
5. Myocardial infarction or acute coronary syndrome within 12 weeks prior to randomization
6. History of malignancy
7. Chronic inflammatory disease that could impact erythropoiesis (for example, systemic lupus erythematosis, rheumatoid arthritis, celiac disease) even if it is currently in remission
8. History of myelodysplastic syndrome, multiple myeloma, or pure red cell aplasia
9. History of hemosiderosis, hemochromatosis or polycystic kidney disease
10. Active hemolysis or diagnosis of hemolytic syndrome
11. Uncontrolled or symptomatic secondary hyperparathyroidism
12. Seizure disorder or receiving anti-epilepsy medication
13. Known bone marrow fibrosis
14. Any prior or scheduled organ transplant
15. Prior treatment with roxadustat or any hypoxia-inducible factor prolyl hydroxylase inhibitor
16. History of alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2010-10-29 (Actual); Primary Completion 2012-06-13 (Actual); Study Completion 2012-06-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (35):
  - Mobile, Alabama
  - Pine Bluff, Arkansas
  - Azusa, California
  - Chula Vista, California
  - Downey, California
  - Northridge, California
  - Paramount, California
  - Riverside, California
  - Whittier, California
  - Yuba City, California
  - Fort Lauderdale, Florida
  - Lauderdale Lakes, Florida
  - Pembroke Pines, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Meridian, Idaho
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Shreveport, Louisiana
  - Bethesda, Maryland
  - Detroit, Michigan
  - Lincoln, Nebraska
  - Mount Laurel, New Jersey
  - Mineola, New York
  - New York, New York
  - Asheville, North Carolina
  - Raleigh, North Carolina
  - Canton, Ohio
  - Orangeburg, South Carolina
  - Knoxville, Tennessee
  - Arlington, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
- Puerto Rico (3):
  - Caguas
  - Ponce
  - San Juan

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Roxadustat Tiered, Weight Based Dosing TIW: Participants received roxadustat capsules, administered orally 3 times weekly (TIW) for 16 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kilograms (kg)], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 60, 100, and 140 milligrams [mg] roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL.
- Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW: Participants received roxadustat capsules orally for 16 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 60, 100, and 140 mg roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants had a dose frequency reduction from TIW to 2 times a week (BIW) at the time of the initial Hb response.
- Cohort C: Roxadustat at 50 mg TIW: Participants received roxadustat capsules at 50 mg, administered orally TIW for 24 weeks. Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 10.5-12 g/dL.
- Cohort D: Roxadustat at 100 mg TIW: Participants received roxadustat capsules at 100 mg, administered orally TIW for 24 weeks. Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 10.5-12 g/dL.
- Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW: Participants received roxadustat capsules for 24 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 70, 100, and 150 mg roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.5 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants had a dose frequency reduction from BIW to 1 time a week (QW) at the time of the initial Hb response.
- Cohort F: Roxadustat at 70 mg BIW Then QW: Participants received roxadustat capsules at 70 mg for 24 weeks. Dose adjustments were implemented (up to a maximum roxadustat dose of 2.5 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants had a dose frequency reduction from TIW to BIW at the time of the initial Hb response. Then after >8 weeks of stable Hb, dose frequency was reduced from BIW to QW.
Period: Overall Study
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Started | 24 | 24 | 24 | 24 | 24 | 25
Safety Population (All participants who received any dose of study drug.) | 24 | 24 | 24 | 24 | 24 | 25
Efficacy Evaluable (EE) Population (All participants who received at least 2 weeks of study drug with a hemoglobin (Hb) Baseline (BL) and a valid post-BL value at 2 weeks into study.) | 23 | 24 | 23 | 24 | 24 | 25
Completed | 21 | 21 | 22 | 23 | 21 | 21
Not Completed | 3 | 3 | 2 | 1 | 3 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 1 | 0 | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Enrolled into the Extension Study | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received any dose of study drug.
Groups:
- Cohort A: Roxadustat Tiered, Weight Based Dosing TIW: Participants received roxadustat capsules, administered orally TIW for 16 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 60, 100, and 140 mg roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL.
- Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW: Participants received roxadustat capsules orally for 16 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 60, 100, and 140 mg roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.2 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants had a dose frequency reduction from TIW to BIW at the time of the initial Hb response.
- Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW: Participants received roxadustat capsules for 24 weeks. Initial roxadustat dose was based on a tiered, weight-based dosing scheme (low-weight [45 to 60 kg], medium-weight [>60 to 90 kg], and heavy-weight [>90 to 140 kg] participants received 70, 100, and 150 mg roxadustat, respectively). Dose adjustments were implemented (up to a maximum roxadustat dose of 2.5 mg/kg per dose) every 4 weeks starting Week 5 to maintain Hb levels at 11-13 g/dL. Participants had a dose frequency reduction from BIW to QW at the time of the initial Hb response.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 25 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.3) | 64.3 (10.3) | 59.2 (14.7) | 69.8 (8.0) | 61.8 (13.2) | 65.2 (8.6) | 64.4 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 16 | 11 | 16 | 13 | 92
  Male | 5 | 7 | 8 | 13 | 8 | 12 | 53
Hb [Mean (Standard Deviation); unit: g/dL] — Baseline was defined as the mean of the last 3 available values predose.
  g/dL | 9.56 (0.86) | 9.67 (0.62) | 9.80 (0.49) | 9.68 (0.77) | 9.89 (0.60) | 9.72 (0.60) | 9.72 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Number (%) of Participants With an Hb Response by Week 17
Description: An Hb response was defined as a Hb level of ≥11 g/dL and an increase from BL ≥1 g/dL.
Time Frame: Up to Week 17
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants | 19 | 24 | 21 | 23 | 23 | 21

2. Secondary Outcome: Number (%) of Participants With an Hb Response by Weeks 5, 9, 13, 17, 21, and 25
Description: An Hb response was defined as a Hb level of ≥11 g/dL and an increase from BL ≥1 g/dL.
Time Frame: Up to Weeks 5, 9, 13, and 17 (all cohorts) and Weeks 21 and 25 (24-week treatment cohorts only)
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants
  Week 5 | 15 | 14 | 3 | 13 | 9 | 9
  Week 9 | 18 | 21 | 12 | 20 | 18 | 13
  Week 13 | 18 | 23 | 15 | 21 | 20 | 16
  Week 17 | 19 | 24 | 17 | 22 | 23 | 20
  Week 21: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Week 21 |  |  | 19 | 22 | 23 | 21
  Week 25: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Week 25 |  |  | 21 | 23 | 23 | 21

3. Secondary Outcome: Change From Baseline in Hb at Weeks 5, 9, 13, 17, 21, and 25
Description: Baseline is defined as the mean of the last 3 available values predose.
Time Frame: Baseline, Weeks 5, 9, 13, and 17 (all cohorts) and Weeks 21 and 25 (24-week treatment cohorts only)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
g/dL
  Baseline | 9.56 (0.88) | 9.67 (0.62) | 9.80 (0.50) | 9.68 (0.77) | 9.89 (0.60) | 9.72 (0.60)
  Change at Week 5: number analyzed (Participants) | 23 | 23 | 23 | 21 | 21 | 24
  Change at Week 5 | 1.71 (1.02) | 1.11 (0.96) | 0.57 (0.65) | 1.65 (0.95) | 0.74 (0.75) | 0.63 (0.85)
  Change at Week 9: number analyzed (Participants) | 21 | 24 | 22 | 20 | 20 | 23
  Change at Week 9 | 2.58 (0.97) | 1.77 (1.18) | 0.99 (0.87) | 2.21 (1.02) | 1.67 (0.98) | 0.89 (1.23)
  Change at Week 13: number analyzed (Participants) | 22 | 23 | 22 | 22 | 22 | 22
  Change at Week 13 | 2.46 (0.93) | 2.06 (1.07) | 1.26 (1.09) | 2.17 (1.19) | 1.43 (0.90) | 1.19 (1.10)
  Change at Week 17: number analyzed (Participants) | 21 | 24 | 22 | 23 | 18 | 20
  Change at Week 17 | 2.63 (0.83) | 2.28 (0.87) | 1.43 (1.15) | 2.26 (1.31) | 1.50 (0.73) | 1.46 (1.23)
  Change at Week 21: number analyzed (Participants) | 0 | 0 | 22 | 21 | 20 | 23
  Change at Week 21 |  |  | 1.30 (0.97) | 1.94 (0.81) | 1.19 (1.08) | 1.79 (0.77)
  Change at Week 25: number analyzed (Participants) | 0 | 0 | 22 | 24 | 20 | 23
  Change at Week 25 |  |  | 1.33 (1.00) | 1.73 (1.14) | 1.28 (1.08) | 1.51 (1.06)

4. Secondary Outcome: Number (%) of Participants With Mean Hb Between 11-12, 11-13, and 10.5-13 g/dL During Weeks 5-8, 9-12, 9-16, 13-16, 17-20, 17-24, 21-24, and 25-28
Description: Participants can have a Hb value reported for more than 1 of the categories (11-12, 11-13, and 10.5-13 g/dL) during the week intervals since these categories are not mutually exclusive.
Time Frame: Weeks 5-8, 9-12, 9-16, 13-16, and 17-20 (all cohorts) and Weeks 17-24, 21-24, and 25-28 (24-week treatment cohorts only)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants
  Weeks 5-8, HB Value of 11-12 g/dL | 4 | 11 | 7 | 8 | 10 | 7
  Weeks 5-8, HB Value of 11-13 g/dL | 13 | 14 | 7 | 12 | 13 | 8
  Weeks 5-8, HB Value of 10.5-13 g/dL | 16 | 18 | 14 | 16 | 17 | 13
  Weeks 9-12, HB Value of 11-12 g/dL | 5 | 12 | 7 | 8 | 9 | 6
  Weeks 9-12, HB Value of 11-13 g/dL | 13 | 18 | 9 | 16 | 12 | 10
  Weeks 9-12, HB Value of 10.5-13 g/dL | 14 | 21 | 16 | 17 | 16 | 15
  Weeks 9-16, HB Value of 11-12 g/dL | 6 | 11 | 8 | 8 | 11 | 7
  Weeks 9-16, HB Value of 11-13 g/dL | 12 | 19 | 11 | 16 | 14 | 11
  Weeks 9-16, HB Value of 10.5-13 g/dL | 14 | 22 | 15 | 19 | 20 | 17
  Weeks 13-16, HB Value of 11-12 g/dL | 6 | 10 | 9 | 9 | 14 | 9
  Weeks 13-16, HB Value of 11-13 g/dL | 11 | 19 | 10 | 17 | 17 | 13
  Weeks 13-16, HB Value of 10.5-13 g/dL | 13 | 21 | 14 | 19 | 20 | 18
  Weeks 17-20, HB Value of 11-12 g/dL | 4 | 9 | 9 | 11 | 9 | 9
  Weeks 17-20, HB Value of 11-13 g/dL | 10 | 18 | 11 | 20 | 11 | 16
  Weeks 17-20, HB Value of 10.5-13 g/dL | 11 | 19 | 17 | 20 | 17 | 19
  Weeks 17-24, HB Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, HB Value of 11-12 g/dL |  |  | 12 | 14 | 11 | 11
  Weeks 17-24, HB Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, HB Value of 11-13 g/dL |  |  | 13 | 20 | 12 | 17
  Weeks 17-24, HB Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, HB Value of 10.5-13 g/dL |  |  | 18 | 22 | 15 | 21
  Weeks 21-24, HB Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, HB Value of 11-12 g/dL |  |  | 11 | 13 | 7 | 14
  Weeks 21-24, HB Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, HB Value of 11-13 g/dL |  |  | 13 | 18 | 9 | 18
  Weeks 21-24, HB Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, HB Value of 10.5-13 g/dL |  |  | 19 | 21 | 13 | 20
  Weeks 25-28, HB Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, HB Value of 11-12 g/dL |  |  | 10 | 8 | 6 | 12
  Weeks 25-28, HB Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, HB Value of 11-13 g/dL |  |  | 11 | 11 | 9 | 13
  Weeks 25-28, HB Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, HB Value of 10.5-13 g/dL |  |  | 16 | 19 | 14 | 17

5. Secondary Outcome: Number (%) of Participants With 2 Consecutive Hb Values Between 11-12, 11-13, and 10.5-13 g/dL During Weeks 5-8, 9-12, 13-16, 9-16, 17-20, 17-24, 21-24, and 25-28
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants
  Weeks 5-8, Hb Value of 11-12 g/dL | 4 | 11 | 5 | 9 | 8 | 4
  Weeks 5-8, Hb Value of 11-13 g/dL | 13 | 14 | 8 | 12 | 12 | 6
  Weeks 5-8, Hb Value of 10.5-13 g/dL | 15 | 17 | 14 | 16 | 16 | 13
  Weeks 9-12, Hb Value of 11-12 g/dL | 5 | 12 | 7 | 8 | 10 | 8
  Weeks 9-12, Hb Value of 11-13 g/dL | 12 | 17 | 10 | 16 | 12 | 11
  Weeks 9-12, Hb Value of 10.5-13 g/dL | 14 | 21 | 16 | 18 | 17 | 15
  Weeks 9-16, Hb Value of 11-12 g/dL | 8 | 16 | 10 | 10 | 15 | 11
  Weeks 9-16, Hb Value of 11-13 g/dL | 14 | 22 | 13 | 20 | 18 | 15
  Weeks 9-16, Hb Value of 10.5-13 g/dL | 16 | 23 | 19 | 20 | 22 | 18
  Weeks 13-16, Hb Value of 11-12 g/dL | 7 | 11 | 9 | 7 | 13 | 7
  Weeks 13-16, Hb Value of 11-13 g/dL | 12 | 19 | 12 | 15 | 17 | 13
  Weeks 13-16, Hb Value of 10.5-13 g/dL | 13 | 20 | 17 | 16 | 20 | 17
  Weeks 17-20, Hb Value of 11-12 g/dL | 0 | 0 | 10 | 10 | 9 | 8
  Weeks 17-20, Hb Value of 11-13 g/dL | 0 | 0 | 12 | 19 | 12 | 14
  Weeks 17-20, Hb Value of 10.5-13 g/dL | 0 | 0 | 16 | 20 | 18 | 20
  Weeks 17-24, Hb Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of 11-12 g/dL |  |  | 14 | 17 | 14 | 17
  Weeks 17-24, Hb Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of 11-13 g/dL |  |  | 16 | 22 | 14 | 20
  Weeks 17-24, Hb Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of 10.5-13 g/dL |  |  | 20 | 22 | 18 | 22
  Weeks 21-24, Hb Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of 11-12 g/dL |  |  | 12 | 12 | 10 | 15
  Weeks 21-24, Hb Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of 11-13 g/dL |  |  | 15 | 18 | 11 | 18
  Weeks 21-24, Hb Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of 10.5-13 g/dL |  |  | 20 | 21 | 14 | 21
  Weeks 25-28, Hb Value of 11-12 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of 11-12 g/dL |  |  | 5 | 9 | 4 | 8
  Weeks 25-28, Hb Value of 11-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of 11-13 g/dL |  |  | 8 | 13 | 7 | 12
  Weeks 25-28, Hb Value of 10.5-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of 10.5-13 g/dL |  |  | 13 | 19 | 14 | 16

6. Secondary Outcome: Number (%) of Participants Who Achieve Maximum Hb Between 11-12, 11-13, and 10.5-13 g/dL by Weeks 5, 9, 13, 17, 21, and 25
Description: Participants can have a Hb value for the same category (11-12, 11-13, or 10.5-13 g/dL) reported for multiple weeks.
Time Frame: Weeks 5, 9, 13, and 17 (all cohorts) and Weeks 21 and 25 (24-week treatment cohorts only)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants
  Hb Value of 11-12 g/dL by Week 5 | 9 | 11 | 5 | 8 | 11 | 10
  Hb Value of 11-12 g/dL by Week 9 | 11 | 16 | 11 | 11 | 15 | 14
  Hb Value of 11-12 g/dL by Week 13 | 11 | 19 | 14 | 13 | 17 | 17
  Hb Value of 11-12 g/dL by Week 17 | 12 | 20 | 16 | 14 | 17 | 20
  Hb Value of 11-12 g/dL by Week 21: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 11-12 g/dL by Week 21 |  |  | 17 | 15 | 19 | 22
  Hb Value of 11-12 g/dL by Week 25: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 11-12 g/dL by Week 25 |  |  | 21 | 18 | 20 | 22
  Hb Value of 11-13 g/dL by Week 5 | 16 | 14 | 6 | 14 | 13 | 10
  Hb Value of 11-13 g/dL by Week 9 | 18 | 21 | 14 | 19 | 18 | 14
  Hb Value of 11-13 g/dL by Week 13 | 18 | 23 | 17 | 21 | 21 | 17
  Hb Value of 11-13 g/dL by Week 17 | 19 | 24 | 19 | 22 | 23 | 21
  Hb Value of 11-13 g/dL by Week 21: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 11-13 g/dL by Week 21 |  |  | 20 | 22 | 23 | 22
  Hb Value of 11-13 g/dL by Week 25: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 11-13 g/dL by Week 25 |  |  | 22 | 23 | 23 | 22
  Hb Value of 10.5-13 g/dL by Week 5 | 17 | 20 | 12 | 17 | 17 | 14
  Hb Value of 10.5-13 g/dL by Week 9 | 19 | 22 | 19 | 21 | 19 | 19
  Hb Value of 10.5-13 g/dL by Week 13 | 19 | 23 | 20 | 23 | 22 | 21
  Hb Value of 10.5-13 g/dL by Week 17 | 20 | 24 | 21 | 23 | 23 | 23
  Hb Value of 10.5-13 g/dL by Week 21: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 10.5-13 g/dL by Week 21 |  |  | 22 | 24 | 23 | 23
  Hb Value of 10.5-13 g/dL by Week 25: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Hb Value of 10.5-13 g/dL by Week 25 |  |  | 23 | 24 | 23 | 24

7. Secondary Outcome: Number (%) of Participants With Maximum Hb <11, >12, >13, and >14 g/dL During Weeks 5-8, 9-12, 9-16, 13-16, 17-20, 17-24, 21-24, and 25-28
Time Frame: as for outcome 4
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
Participants
  Weeks 5-8, Hb Value of <11 g/dL | 6 | 9 | 10 | 5 | 6 | 13
  Weeks 5-8, Hb Value of 12-13 g/dL | 10 | 6 | 4 | 6 | 4 | 3
  Weeks 5-8, Hb Value of 13-14 g/dL | 2 | 1 | 0 | 3 | 1 | 0
  Weeks 5-8, Hb Value of >14 g/dL | 1 | 0 | 0 | 1 | 0 | 0
  Weeks 9-12, Hb Value of <11 g/dL | 4 | 2 | 9 | 4 | 7 | 11
  Weeks 9-12, Hb Value of 12-13 g/dL | 5 | 9 | 4 | 8 | 6 | 6
  Weeks 9-12, Hb Value of 13-14 g/dL | 7 | 1 | 1 | 3 | 3 | 0
  Weeks 9-12, Hb Value of >14 g/dL | 2 | 1 | 0 | 2 | 0 | 0
  Weeks 9-16, Hb Value of <11 g/dL | 4 | 1 | 7 | 1 | 2 | 7
  Weeks 9-16, Hb Value of 12-13 g/dL | 4 | 10 | 5 | 8 | 9 | 8
  Weeks 9-16, Hb Value of 13-14 g/dL | 7 | 4 | 2 | 6 | 3 | 1
  Weeks 9-16, Hb Value of >14 g/dL | 4 | 1 | 0 | 3 | 0 | 0
  Weeks 13-16, Hb Value of <11 g/dL | 5 | 2 | 9 | 1 | 3 | 7
  Weeks 13-16, Hb Value of 12-13 g/dL | 4 | 9 | 4 | 8 | 7 | 7
  Weeks 13-16, Hb Value of 13-14 g/dL | 6 | 4 | 2 | 7 | 3 | 1
  Weeks 13-16, Hb Value of >14 g/dL | 2 | 0 | 0 | 1 | 0 | 0
  Weeks 17-20, Hb Value of <11 g/dL | 4 | 3 | 5 | 2 | 3 | 4
  Weeks 17-20, Hb Value of 12-13 g/dL | 6 | 9 | 4 | 10 | 5 | 5
  Weeks 17-20, Hb Value of 13-14 g/dL | 6 | 3 | 1 | 6 | 0 | 2
  Weeks 17-20, Hb Value of >14 g/dL | 1 | 0 | 0 | 0 | 1 | 0
  Weeks 17-24, Hb Value of <11 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of <11 g/dL |  |  | 2 | 0 | 3 | 3
  Weeks 17-24, Hb Value of 12-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of 12-13 g/dL |  |  | 8 | 13 | 6 | 7
  Weeks 17-24, Hb Value of 13-14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of 13-14 g/dL |  |  | 1 | 6 | 0 | 4
  Weeks 17-24, Hb Value of >14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 17-24, Hb Value of >14 g/dL |  |  | 0 | 0 | 1 | 0
  Weeks 21-24, Hb Value of <11 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of <11 g/dL |  |  | 2 | 1 | 9 | 4
  Weeks 21-24, Hb Value of 12-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of 12-13 g/dL |  |  | 6 | 10 | 3 | 7
  Weeks 21-24, Hb Value of 13-14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of 13-14 g/dL |  |  | 1 | 1 | 1 | 3
  Weeks 21-24, Hb Value of >14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 21-24, Hb Value of >14 g/dL |  |  | 0 | 0 | 0 | 0
  Weeks 25-28, Hb Value of <11 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of <11 g/dL |  |  | 7 | 6 | 7 | 8
  Weeks 25-28, Hb Value of 12-13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of 12-13 g/dL |  |  | 4 | 4 | 4 | 3
  Weeks 25-28, Hb Value of 13-14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of 13-14 g/dL |  |  | 0 | 1 | 0 | 1
  Weeks 25-28, Hb Value of >14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 24 | 24 | 25
  Weeks 25-28, Hb Value of >14 g/dL |  |  | 0 | 0 | 0 | 0

8. Secondary Outcome: Median Time to Hb Response: Hb Increase ≥1 g/dL From Baseline and Hb ≥11 g/dL
Description: Median time to response was estimated using Kaplan Meier method, Cohort A and B censored at Week 17, Cohort C, D, E, and F censored at Week 25. The median number of days presented was calculated from Baseline to the day the Hb response was achieved.
Time Frame: Up to Week 17 (Cohorts A and B) and up to Week 25 (Cohorts C-F)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
days | 28.0 [28.0 to 56.0] | 28.0 [28.0 to 56.0] | 48.9 [28.0 to 56.0] | 28.0 [28.0 to 56.0] | 35.0 [28.0 to 56.0] | 56.0 [28.0 to 56.0]

9. Secondary Outcome: Median Initial Hb Responsive Time: Time to Initial Hb Increase ≥1.0 g/dL From Baseline
Description: Median time to response was estimated using Kaplan Meier method; Cohort A and B censored at Week 17 and Cohort C, D, E, and F censored at Week 25. The median number of days presented was calculated from Baseline to the day the Hb response was achieved.
Time Frame: Up to Week 17 (Cohorts A and B) and up to Week 25 (Cohorts C, D, E, and F)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
days | 21.0 [21.0 to 42.0] | 21.6 [21.0 to 42.0] | 42.0 [21.0 to 42.0] | 21.0 [21.0 to 42.0] | 35.0 [21.0 to 42.0] | 42.0 [21.0 to 42.0]

10. Secondary Outcome: Median Initial Hb Responsive Dose: Dose at Which Initial Hb Increases to ≥1.0 g/dL From Baseline
Time Frame: Up to Week 17 (Cohorts A and B) and up to Week 25 (Cohorts C-F)
Population: as for outcome 1
Measure: Median (Full Range); unit: mg/kg/week
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 25
mg/kg/week | 2.30 [0.6 to 6.4] | 2.50 [1.4 to 4.4] | 2.32 [0.7 to 6.6] | 2.36 [0.8 to 6.5] | 1.96 [0.5 to 4.9] | 1.61 [0.8 to 4.6]

11. Secondary Outcome: Change in Hb After Reaching a Hb Response of ≥11.0 g/dL and an Increase in Hb by ≥1.0 g/dL by Week
Time Frame: Cohorts A and B: Weekly through Week 16 (end of treatment), Week 18 (2 weeks posttreatment), and Week 20 (4 weeks posttreatment); Cohorts C-F: Weekly through Week 24 (end of treatment), Week 26 (2 weeks posttreatment), and Week 28 (4 weeks posttreatment)
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 19 | 24 | 21 | 23 | 23 | 21
g/dL
  Hb at Response Timepoint | 11.49 (0.414) | 11.40 (0.289) | 11.32 (0.360) | 11.47 (0.430) | 11.62 (0.543) | 11.43 (0.348)
  Change after 1 week: number analyzed (Participants) | 17 | 23 | 21 | 22 | 23 | 19
  Change after 1 week | 0.30 (0.579) | 0.03 (0.562) | -0.18 (0.854) | 0.18 (0.570) | -0.26 (0.709) | -0.23 (0.394)
  Change after 2 weeks: number analyzed (Participants) | 18 | 23 | 20 | 23 | 22 | 19
  Change after 2 weeks | 0.46 (0.685) | 0.05 (0.634) | -0.22 (0.868) | 0.41 (0.678) | -0.34 (0.720) | -0.21 (0.707)
  Change after 3 weeks: number analyzed (Participants) | 17 | 21 | 19 | 23 | 23 | 19
  Change after 3 weeks | 0.67 (0.635) | 0.19 (0.720) | -0.02 (0.842) | 0.44 (0.873) | -0.31 (0.934) | -0.25 (0.682)
  Change after 4 weeks: number analyzed (Participants) | 18 | 23 | 19 | 22 | 23 | 18
  Change after 4 weeks | 0.81 (0.642) | 0.17 (0.968) | 0.06 (0.767) | 0.61 (0.859) | -0.18 (1.080) | -0.24 (0.794)
  Change after 5 weeks: number analyzed (Participants) | 17 | 23 | 18 | 19 | 23 | 19
  Change after 5 weeks | 0.99 (0.705) | 0.20 (1.004) | -0.07 (0.701) | 0.65 (0.883) | -0.05 (1.295) | 0.13 (0.752)
  Change after 6 weeks: number analyzed (Participants) | 18 | 23 | 18 | 21 | 21 | 19
  Change after 6 weeks | 1.01 (0.999) | 0.23 (0.931) | 0.02 (0.821) | 0.67 (0.799) | 0.10 (1.274) | -0.01 (0.937)
  Change after 7 weeks: number analyzed (Participants) | 18 | 23 | 18 | 22 | 22 | 19
  Change after 7 weeks | 0.97 (0.874) | 0.21 (0.860) | 0.40 (0.876) | 0.87 (0.882) | -0.21 (1.255) | 0.03 (0.830)
  Change after 8 weeks: number analyzed (Participants) | 18 | 21 | 16 | 22 | 22 | 20
  Change after 8 weeks | 1.05 (0.852) | 0.45 (0.827) | 0.18 (0.820) | 0.78 (0.820) | -0.15 (1.238) | -0.03 (1.005)
  Change after 9 weeks: number analyzed (Participants) | 17 | 18 | 15 | 22 | 23 | 18
  Change after 9 weeks | 0.88 (0.904) | 0.59 (0.898) | 0.22 (1.131) | 0.79 (0.960) | -0.43 (1.075) | -0.03 (0.944)
  Change after 10 weeks: number analyzed (Participants) | 17 | 14 | 14 | 20 | 22 | 17
  Change after 10 weeks | 0.88 (1.044) | 0.68 (0.787) | 0.44 (1.109) | 1.01 (0.629) | -0.22 (1.226) | 0.26 (1.018)
  Change after 11 weeks: number analyzed (Participants) | 16 | 14 | 15 | 22 | 19 | 16
  Change after 11 weeks | 0.89 (1.088) | 0.59 (0.644) | 0.39 (0.972) | 0.82 (0.678) | -0.42 (0.966) | 0.09 (0.974)
  Change after 12 weeks: number analyzed (Participants) | 15 | 12 | 15 | 21 | 18 | 16
  Change after 12 weeks | 0.91 (1.007) | 0.69 (0.474) | 0.25 (0.966) | 0.60 (0.745) | -0.38 (0.818) | 0.21 (0.774)
  Change after 13 weeks: number analyzed (Participants) | 8 | 7 | 14 | 20 | 16 | 15
  Change after 13 weeks | 1.53 (0.962) | 0.90 (0.837) | 0.13 (1.010) | 0.45 (0.808) | -0.58 (0.946) | 0.33 (0.880)
  Change after 14 weeks: number analyzed (Participants) | 5 | 5 | 14 | 19 | 17 | 15
  Change after 14 weeks | 2.16 (0.385) | 0.94 (0.976) | 0.18 (0.913) | 0.37 (0.874) | -0.65 (1.079) | 0.41 (0.778)
  Change after 15 weeks: number analyzed (Participants) | 1 | 1 | 12 | 19 | 16 | 13
  Change after 15 weeks | 1.20 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 1.50 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 0.13 (0.751) | 0.32 (0.815) | -0.67 (1.191) | 0.18 (0.636)
  Change after 16 weeks: number analyzed (Participants) | 0 | 0 | 11 | 19 | 14 | 13
  Change after 16 weeks |  |  | 0.08 (0.851) | 0.21 (0.808) | -0.68 (1.262) | 0.41 (0.524)
  Change after 17 weeks: number analyzed (Participants) | 0 | 0 | 11 | 19 | 13 | 11
  Change after 17 weeks |  |  | 0.12 (0.529) | 0.18 (0.718) | -0.52 (0.984) | 0.47 (0.751)
  Change after 18 weeks: number analyzed (Participants) | 0 | 0 | 10 | 16 | 12 | 11
  Change after 18 weeks |  |  | -0.06 (0.704) | 0.39 (0.763) | -0.44 (0.699) | 0.27 (0.405)
  Change after 19 weeks: number analyzed (Participants) | 0 | 0 | 6 | 15 | 10 | 10
  Change after 19 weeks |  |  | -0.20 (0.807) | 0.33 (0.855) | -0.31 (0.888) | 0.26 (0.821)
  Change after 20 weeks: number analyzed (Participants) | 0 | 0 | 2 | 13 | 7 | 9
  Change after 20 weeks |  |  | -0.50 (0.283) | -0.12 (1.035) | -0.43 (1.275) | 0.51 (0.839)
  Change after 21 weeks: number analyzed (Participants) | 0 | 0 | 1 | 8 | 4 | 6
  Change after 21 weeks |  |  | 0.20 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -0.49 (1.146) | -0.40 (0.849) | 0.37 (0.737)
  Change after 22 weeks: number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 2
  Change after 22 weeks |  |  | 0.90 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -1.05 (0.480) | -0.33 (0.839) | 0.15 (0.354)
  Change after 23 weeks: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0
  Change after 23 weeks |  |  |  | -1.10 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | -0.90 (NA) — NA=Standard Deviation cannot be calculated with N of 1. |
  Change after 2 weeks posttreatment: number analyzed (Participants) | 19 | 20 | 18 | 22 | 19 | 19
  Change after 2 weeks posttreatment | 0.49 (1.113) | 0.21 (0.985) | -0.28 (0.614) | -0.25 (0.924) | -0.61 (1.023) | -0.34 (0.562)
  Change after 4 weeks posttreatment: number analyzed (Participants) | 19 | 21 | 21 | 22 | 20 | 18
  Change after 4 weeks posttreatment | 0.21 (1.289) | -0.28 (0.902) | -0.62 (0.846) | -0.80 (0.708) | -0.99 (1.296) | -0.79 (0.777)

12. Secondary Outcome: Mean Hb Values From Participants Who Reached Hb >11.0 g/dL in the Hb 11-12, 11-13, and 10.5-13 g/dL Categories
Time Frame: Cohorts A and B: Weekly through Week 16 (end of treatment [EoT]) and Week 20 (Follow up [4 weeks posttreatment]); Cohorts C-F: Weekly through Week 24 (EoT) and Week 28 (Follow up [4 weeks posttreatment])
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 19 | 23 | 22 | 23 | 23 | 22
g/dL
  After Response through EoT, Hb Category <11 g/dL | 11.50 (25.937) | 18.75 (27.254) | 35.48 (32.727) | 14.03 (18.311) | 38.32 (30.175) | 32.56 (33.384)
  After Response through EoT, Hb Category 11-12 g/dL | 31.46 (30.410) | 48.86 (26.771) | 46.67 (29.540) | 41.54 (26.619) | 44.17 (22.858) | 47.00 (27.692)
  After Response through EoT, Hb Category 11-13 g/dL | 66.73 (27.453) | 76.05 (26.577) | 62.10 (31.528) | 74.96 (24.078) | 56.92 (27.338) | 64.39 (32.083)
  After Response through EoT, Hb Category 10.5-13 g/dL | 76.80 (23.899) | 87.20 (20.118) | 82.69 (25.854) | 83.50 (21.354) | 79.01 (23.045) | 83.97 (26.219)
  In Follow Up, Hb Category <11 g/dL: number analyzed (Participants) | 18 | 21 | 21 | 23 | 20 | 19
  In Follow Up, Hb Category <11 g/dL | 16.67 (34.300) | 35.71 (42.258) | 54.76 (41.547) | 47.83 (43.896) | 57.50 (43.755) | 50.00 (44.096)
  In Follow Up, Hb Category 11-12 g/dL: number analyzed (Participants) | 18 | 21 | 21 | 23 | 20 | 19
  In Follow Up, Hb Category 11-12 g/dL | 30.56 (38.877) | 40.48 (40.679) | 40.48 (40.679) | 41.30 (38.883) | 30.00 (37.697) | 47.37 (42.406)
  In Follow Up, Hb Category 11-13 g/dL: number analyzed (Participants) | 18 | 21 | 21 | 23 | 20 | 19
  In Follow Up, Hb Category 11-13 g/dL | 69.44 (42.492) | 59.52 (40.679) | 45.24 (41.547) | 52.17 (43.896) | 42.50 (43.755) | 50.00 (44.096)
  In Follow Up, Hb Category 10.5-13 g/dL: number analyzed (Participants) | 18 | 21 | 21 | 23 | 20 | 19
  In Follow Up, Hb Category 10.5-13 g/dL | 75.00 (39.295) | 83.33 (32.914) | 66.67 (36.515) | 71.74 (39.388) | 65.00 (43.225) | 73.68 (34.835)

13. Secondary Outcome: Mean of Weekly Hb Values <10.5, >13, and >14 g/dL During Weeks 13-17 and 18-25
Description: The mean percentage of the scheduled weekly Hb values that were <10.5, >13, and >14 g/dL during Weeks 13-17 and 18-25 is presented.
Time Frame: Weeks 13-17 (all cohorts) and 18-25 (24-week treatment cohorts only)
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: percentage of Hb values
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 22 | 24 | 23 | 23 | 22 | 24
percentage of Hb values
  Weeks 13-17, Hb <10.5 g/dL: number analyzed (Participants) | 22 | 24 | 23 | 23 | 22 | 23
  Weeks 13-17, Hb <10.5 g/dL | 15.23 (33.893) | 7.92 (20.212) | 25.65 (36.752) | 9.78 (24.885) | 9.17 (19.174) | 22.75 (35.995)
  Weeks 13-17, Hb >13 g/dL: number analyzed (Participants) | 22 | 24 | 23 | 23 | 22 | 23
  Weeks 13-17, Hb >13 g/dL | 25.00 (37.257) | 7.50 (17.508) | 4.35 (14.717) | 18.26 (31.283) | 2.95 (7.662) | 0.87 (4.170)
  Weeks 13-17, Hb >14 g/dL: number analyzed (Participants) | 22 | 24 | 23 | 23 | 22 | 23
  Weeks 13-17, Hb >14 g/dL | 2.73 (9.351) | 0 (0) | 0 (0) | 0.87 (4.170) | 0 (0) | 0 (0)
  Weeks 18-25, Hb <10.5 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 23 | 22 | 24
  Weeks 18-25, Hb <10.5 g/dL |  |  | 21.97 (31.809) | 9.38 (22.797) | 23.86 (33.830) | 16.84 (31.625)
  Weeks 18-25, Hb >13 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 23 | 22 | 24
  Weeks 18-25, Hb >13 g/dL |  |  | 2.17 (10.426) | 5.00 (16.219) | 3.41 (15.990) | 3.13 (7.599)
  Weeks 18-25, Hb >14 g/dL: number analyzed (Participants) | 0 | 0 | 23 | 23 | 22 | 24
  Weeks 18-25, Hb >14 g/dL |  |  | 0 (0) | 0 (0) | 0.57 (2.665) | 0 (0)

14. Secondary Outcome: Number (%) of Participants Requiring Rescue Therapy
Description: Rescue treatment included recombinant erythropoiesis-stimulating agent (ESA), red blood cell transfusion (in the absence of a known bleeding episode or surgical blood loss), or intravenous (IV) Iron
Time Frame: Baseline up to Week 28 (end of study)
Population: Safety Population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 25
Participants
  Blood Transfusion | 0 | 2 | 0 | 1 | 2 | 0
  ESA | 0 | 1 | 0 | 0 | 1 | 2
  IV Iron | 0 | 1 | 0 | 1 | 2 | 2

15. Secondary Outcome: Number (%) of Participants Requiring Therapeutic Phlebotomy
Time Frame: Baseline up to Week 28 (end of study)
Population: Safety Population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 25
Participants | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number (%) of Participants Withdrawn From the Study Due to Inadequate Efficacy
Time Frame: Baseline up to Week 28 (end of study)
Population: Safety Population included all participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 25
Participants | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number (%) of Participants With Dose Changes During Weeks 1-4, 5-12, 13-16, and 17-24
Description: Dose changes include dose reductions, dose increases, and dose holds.
Time Frame: Weeks 1-4, 5-12, and 13-16 (all cohorts) and Weeks 17-24 (24-week treatment cohorts only)
Population: Safety Population included all participants who received any dose of study drug. Here, 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 25
Participants
  Dose reduced, Weeks 1-4 | 5 | 1 | 0 | 2 | 1 | 0
  Dose reduced, Weeks 5-12 | 13 | 4 | 2 | 7 | 3 | 5
  Dose reduced, Weeks 13-16 | 0 | 7 | 4 | 3 | 1 | 0
  Dose reduced, Weeks 17-24: number analyzed (Participants) | 0 | 0 | 24 | 24 | 24 | 25
  Dose reduced, Weeks 17-24 |  |  | 2 | 3 | 1 | 2
  Dose increased, Weeks 1-4 | 0 | 0 | 0 | 0 | 0 | 0
  Dose increased, Weeks 5-12 | 10 | 11 | 14 | 9 | 9 | 15
  Dose increased, Weeks 13-16 | 4 | 4 | 2 | 1 | 3 | 4
  Dose increased, Weeks 17-24: number analyzed (Participants) | 0 | 0 | 24 | 24 | 24 | 25
  Dose increased, Weeks 17-24 |  |  | 2 | 3 | 5 | 0
  Dose held, Weeks 1-4 | 2 | 4 | 0 | 2 | 3 | 3
  Dose held, Weeks 5-12 | 5 | 2 | 2 | 4 | 3 | 4
  Dose held, Weeks 13-16 | 1 | 1 | 0 | 1 | 2 | 0
  Dose held, Weeks 17-24: number analyzed (Participants) | 0 | 0 | 24 | 24 | 24 | 25
  Dose held, Weeks 17-24 |  |  | 1 | 1 | 3 | 0

18. Secondary Outcome: Weekly Total Dose and Cumulative Total Dose (mg/kg) When First Achieving Hb Response (Hb Increase ≥1 g/dL From Baseline and Hb ≥11 g/dL)
Time Frame: Cohorts A and B: Weekly through Week 16 (end of treatment); Cohorts C-F: Weekly through Week 24 (end of treatment)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 19 | 24 | 21 | 23 | 23 | 21
mg/kg
  Weekly Dose | 4.08 (0.952) | 4.13 (0.944) | 2.88 (1.721) | 4.17 (1.119) | 2.65 (0.886) | 3.02 (0.876)
  Cumulative Dose | 16.86 (17.097) | 20.05 (15.994) | 24.41 (23.838) | 21.21 (18.229) | 16.57 (12.154) | 22.16 (17.612)

19. Secondary Outcome: Mean Weekly Dose After Achieving First Hb Response (Hb Increase ≥1 g/dL From Baseline and Hb ≥11 g/dL)
Time Frame: Cohorts A and B: Weekly through Week 16 (end of treatment); Cohorts C-F: Weekly through Week 24 (end of treatment)
Population: Safety Population included all participants who received any dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 18 | 23 | 20 | 23 | 22 | 20
mg/kg
  1 week after response: number analyzed (Participants) | 18 | 23 | 20 | 23 | 22 | 19
  1 week after response | 2.99 (1.16) | 3.05 (1.13) | 2.73 (1.56) | 3.87 (1.28) | 2.09 (0.89) | 2.59 (0.90)
  2 weeks after response: number analyzed (Participants) | 18 | 23 | 19 | 23 | 22 | 20
  2 weeks after response | 2.64 (1.14) | 2.86 (1.13) | 2.63 (1.39) | 3.85 (1.08) | 1.97 (0.92) | 2.50 (1.02)
  3 weeks after response: number analyzed (Participants) | 17 | 21 | 19 | 22 | 22 | 20
  3 weeks after response | 2.50 (0.84) | 2.86 (1.06) | 2.63 (1.39) | 3.53 (1.13) | 1.92 (0.87) | 2.47 (0.99)
  4 weeks after response: number analyzed (Participants) | 18 | 23 | 18 | 22 | 22 | 20
  4 weeks after response | 2.18 (0.82) | 2.82 (0.91) | 2.44 (1.13) | 3.81 (1.36) | 1.96 (0.95) | 2.62 (1.14)
  5 weeks after response: number analyzed (Participants) | 17 | 23 | 18 | 22 | 21 | 18
  5 weeks after response | 2.32 (0.75) | 2.73 (0.86) | 2.54 (1.52) | 3.61 (1.49) | 1.97 (0.96) | 2.57 (1.05)
  6 weeks after response: number analyzed (Participants) | 18 | 22 | 18 | 20 | 20 | 19
  6 weeks after response | 2.09 (0.82) | 2.75 (0.87) | 2.57 (1.47) | 3.48 (1.30) | 1.99 (0.98) | 2.53 (1.16)
  7 weeks after response: number analyzed (Participants) | 17 | 20 | 17 | 21 | 19 | 19
  7 weeks after response | 2.03 (0.69) | 2.76 (0.90) | 2.65 (1.51) | 3.31 (1.29) | 1.99 (1.00) | 2.33 (0.94)
  8 weeks after response: number analyzed (Participants) | 16 | 17 | 16 | 21 | 19 | 19
  8 weeks after response | 2.01 (0.78) | 2.84 (0.96) | 2.60 (1.54) | 3.21 (1.33) | 2.07 (1.07) | 2.14 (0.80)
  9 weeks after response: number analyzed (Participants) | 16 | 15 | 15 | 20 | 18 | 18
  9 weeks after response | 2.01 (0.88) | 2.71 (1.08) | 2.35 (1.22) | 3.16 (1.43) | 2.15 (1.08) | 2.23 (0.86)
  10 weeks after response: number analyzed (Participants) | 15 | 13 | 15 | 20 | 18 | 16
  10 weeks after response | 2.15 (0.79) | 2.59 (1.00) | 2.18 (1.29) | 2.96 (1.36) | 2.13 (1.09) | 2.16 (0.89)
  11 weeks after response: number analyzed (Participants) | 13 | 12 | 15 | 19 | 16 | 15
  11 weeks after response | 2.13 (0.85) | 2.72 (1.16) | 2.18 (1.29) | 2.77 (1.30) | 2.02 (0.89) | 2.14 (0.93)
  12 weeks after response: number analyzed (Participants) | 8 | 5 | 14 | 19 | 16 | 15
  12 weeks after response | 2.07 (0.75) | 2.81 (0.97) | 2.19 (1.34) | 2.65 (1.40) | 1.89 (0.93) | 1.87 (0.82)
  13 weeks after response: number analyzed (Participants) | 4 | 3 | 14 | 19 | 17 | 14
  13 weeks after response | 1.72 (0.85) | 2.70 (0.43) | 2.19 (1.34) | 2.65 (1.42) | 1.70 (0.58) | 1.95 (0.83)
  14 weeks after response: number analyzed (Participants) | 0 | 1 | 13 | 19 | 16 | 14
  14 weeks after response |  | 2.87 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 2.04 (1.42) | 2.69 (1.52) | 1.71 (0.54) | 1.83 (0.87)
  15 weeks after response: number analyzed (Participants) | 0 | 0 | 12 | 19 | 15 | 13
  15 weeks after response |  |  | 2.04 (1.44) | 2.68 (1.51) | 1.70 (0.56) | 1.85 (0.91)
  16 weeks after response: number analyzed (Participants) | 0 | 0 | 12 | 18 | 13 | 11
  16 weeks after response |  |  | 2.04 (1.44) | 2.72 (1.62) | 1.66 (0.53) | 1.76 (0.72)
  17 weeks after response: number analyzed (Participants) | 0 | 0 | 11 | 16 | 13 | 11
  17 weeks after response |  |  | 2.13 (1.46) | 2.51 (1.67) | 1.66 (0.50) | 1.82 (0.89)
  18 weeks after response: number analyzed (Participants) | 0 | 0 | 6 | 14 | 10 | 10
  18 weeks after response |  |  | 1.53 (0.66) | 2.43 (1.79) | 1.57 (0.50) | 1.83 (0.94)
  19 weeks after response: number analyzed (Participants) | 0 | 0 | 3 | 12 | 7 | 9
  19 weeks after response |  |  | 1.25 (0.39) | 2.51 (1.94) | 1.63 (0.58) | 1.89 (0.98)
  20 weeks after response: number analyzed (Participants) | 0 | 0 | 0 | 8 | 4 | 6
  20 weeks after response |  |  |  | 1.82 (1.29) | 1.49 (0.70) | 1.36 (0.40)
  21 weeks after response: number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 2
  21 weeks after response |  |  | 1.65 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 1.13 (0.42) | 1.36 (0.80) | 1.28 (0.24)
  22 weeks after response: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0
  22 weeks after response |  |  |  | 0.85 (NA) — NA=Standard Deviation cannot be calculated with N of 1. | 2.04 (NA) — NA=Standard Deviation cannot be calculated with N of 1. |

20. Secondary Outcome: Change From Baseline in Hb Stratified by Baseline Ferritin >100 Nanograms/Milliliter (ng/mL) and Transferrin Saturation >20% at Week 16 and Week 24
Description: Baseline was defined as the mean of the last 3 available values predose.
Time Frame: Baseline, Weeks 16 (Cohorts A and B End of Treatment) and Week 24 (Cohorts C-F End of Treatment)
Population: EE Population included all participants who received at least 2 weeks of study drug with a Hb BL and a valid post-BL value at 2 weeks into study. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at the specified timepoint. Last-observation-carried-forward (LOCF) method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Number analyzed (Participants) | 17 | 11 | 10 | 14 | 9 | 13
g/dL
  Baseline | 9.62 (0.92) | 9.56 (0.43) | 9.68 (0.41) | 9.58 (0.86) | 9.96 (0.51) | 9.75 (0.63)
  Change at Week 16 | 2.42 (1.12) | 2.32 (1.00) | 1.85 (1.34) | 2.21 (1.42) | 1.37 (0.68) | 1.42 (1.01)
  Change at Week 24: number analyzed (Participants) | 0 | 0 | 10 | 14 | 9 | 13
  Change at Week 24 |  |  | 1.66 (0.45) | 1.75 (1.14) | 1.09 (0.82) | 1.53 (0.88)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 28 (end of study)
Description: Safety Population included all participants who received any dose of study drug.
Arm/Group | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW | Cohort C: Roxadustat at 50 mg TIW | Cohort D: Roxadustat at 100 mg TIW | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW | Cohort F: Roxadustat at 70 mg BIW Then QW
Serious Adverse Events (participants affected / at risk) | 3/24 | 4/24 | 4/24 | 4/24 | 10/24 | 10/25
Other Adverse Events (participants affected / at risk) | 15/24 | 15/24 | 10/24 | 10/24 | 11/24 | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW (N=24) | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW (N=24) | Cohort C: Roxadustat at 50 mg TIW (N=24) | Cohort D: Roxadustat at 100 mg TIW (N=24) | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW (N=24) | Cohort F: Roxadustat at 70 mg BIW Then QW (N=25)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 3
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 1
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diabetic Gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperglycaemic Hyperosmolar Nonketotic Syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Brain Stem Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cerebellar Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Foreign Body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Roxadustat Tiered, Weight Based Dosing TIW (N=24) | Cohort B: Roxadustat Tiered, Weight Based Dosing TIW Then BIW (N=24) | Cohort C: Roxadustat at 50 mg TIW (N=24) | Cohort D: Roxadustat at 100 mg TIW (N=24) | Cohort E: Roxadustat Tiered, Weight Based Dosing BIW Then QW (N=24) | Cohort F: Roxadustat at 70 mg BIW Then QW (N=25)
Urinary Tract Infection (Infections and infestations) | 0 | 4 | 2 | 1 | 4 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2 | 2 | 2 | 3 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 2 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 1 | 3 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 2 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 2 | 2 | 0
Oedema Peripheral (General disorders) | 1 | 5 | 4 | 2 | 2 | 4
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 1 | 2 | 0
Headache (Nervous system disorders) | 3 | 1 | 1 | 2 | 0 | 1
Hypertension (Vascular disorders) | 4 | 1 | 1 | 2 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other